CLINICAL TRIAL: NCT03939637
Title: A Phase III Study of Eltrombopag vs Standard Front Line Management for Newly Diagnosed Immune Thrombocytopenia in Children
Brief Title: Eltrombopag vs Standard Front Line Management for Newly Diagnosed Immune Thrombocytopenia (ITP) in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Boston Children's Hospital (Other); University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Amanda Grimes, Assistant Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-42131 ICON 3; CETB115JUS33T (Other: Novartis); ICON 3 (Other: ICON Consortium)
Record Dates: First submitted 2019-04-25; First posted 2019-05-07 (Actual); Results first posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Immune Thrombocytopenia
Keywords: ITP; Immune Thrombocytopenia; Newly Diagnosed Immune Thrombocytopenia; Newly Diagnosed ITP
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — eltrombopag; Steroids; Immunoglobulins, Intravenous; Rho(D) Immune Globulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Eltrombopag (Experimental): Patients randomized to eltrombopag will be treated for 12 weeks, with the possibility to continue therapy for up to 1 year depending on response.
  Interventions: Drug: Eltrombopag
- Standard first-line therapy (Active Comparator): Subjects randomized to the standard therapy arm will receive one of three treatments at the discretion of the treating physician. Patients who previously failed standard management prior to study entry must be treated with a different agent than their original failed agent. e.g. Patient who failed steroids could receive either IVIg or anti-D if randomized to the standard treatment arm.
  Standard therapy will be administered as commercially available drug.
  Investigator may choose amongst the following:
  * IVIg: IVIG 1 g/kg x1 (no steroids for pre-medication or adjunctive therapy)
  * Steroids: Prednisone/Prednisolone 4 mg/kg/day (Max 120 mg/day) x 4 days
  * Rho(D) Immune Globulin: Anti-D globulin 75 mcg/kg x1 (no steroids for pre-medication or adjunctive therapy)
  Interventions: Drug: Steroids; Drug: IVIG; Drug: Rho(D) Immune Globulin

INTERVENTIONS:
Drug: Eltrombopag — Starting dose for eltrombopag will be based on manufacturer recommendations, and drug will be titrated to effect per guidelines.
  * Children 1 to 5 years: Initial: 25 mg once daily
  * Children ≥6 years and Adolescents: Initial: 50 mg once daily (25 mg once daily for patients of East-Asian ethnicity [e.g., Chinese, Japanese, Korean, Taiwanese])
  Dose should be titrated based on platelet response. Maximum dose: 75 mg once daily.
  Arms: Eltrombopag
Drug: Steroids — Prednisone/Prednisolone 4mg/kg/day (Max 120 mg/day) x 4 day
  Arms: Standard first-line therapy
Drug: IVIG — IVIG 1 g/kg x1 (no steroids for pre-medication or adjunctive therapy)
  Arms: Standard first-line therapy
Drug: Rho(D) Immune Globulin — Anti-D globulin 75 mcg/kg x1 (no steroids for pre-medication or adjunctive therapy)
  Arms: Standard first-line therapy

SUMMARY:
This is an investigator initiated, multicenter, open label, randomized phase 3 study for subjects with newly diagnosed ITP from ages 1 to less than 18 years old.

DETAILED DESCRIPTION:
This is a prospective, open label, randomized, two-arm, multi-center Phase 3 trial.

Patients with newly diagnosed ITP are randomized 2:1 to receive the experimental treatment, eltrombopag, or investigator's choice of 3 standard therapies. The primary objective is to determine if the proportion of patients with platelet response is significantly greater in patients treated with eltrombopag compared to those treated with standard therapies.

ELIGIBILITY:
Inclusion Criteria:

* Age: 1- <18 years
* Newly diagnosed ITP (<3 months from diagnosis (first abnormal platelet count), per international working group definition17)
* Platelets <30 x 10^9/L at screening
* Requires pharmacologic treatment from the perspective of the treating clinician.

Need to treat is at the discretion of the investigator, but there should be clinical equipoise about the use of eltrombopag vs standard treatment options (patients should not, in the opinion of the investigator, require concomitant therapy at time of enrollment).

* Treatment options include one of three standard therapies, (IVIg, steroids, or Anti-D). For example, if patient has previously shown no response to IVIg or steroids and is Rh-negative, patient would not be eligible for study.
* Patient population includes both:

  1. Upfront treatment: Patient within 10 days of ITP diagnosis who has not received previous treatment OR
  2. Treatment failure: Patients who have failed standard management (observation or treatment with one or more first-line agents)

     * Failure of observation: no platelet recovery (>30 x 10^9/L) with observation >10 days from diagnosis, with need to treat
     * Poor response to first-line agent (platelets remain <30 x10^9/L)
     * Initial response to first-line agent, but response wanes and platelets fall below 30 x10^9/L
* Family willing and able to return for required lab studies

Exclusion Criteria:

* Severe bleeding: Buchanan Overall Grade 4 or 5 bleeding, or severe bleeding requiring emergent treatment at the discretion of the provider. (e.g., intracranial hemorrhage, pulmonary hemorrhage, bleeding with ongoing need for pRBC transfusion)
* Prior treatment with TPO-RA (eltrombopag or romiplostim)
* Known secondary ITP (due to lupus, CVID, ALPS)
* Known HIV (or history of HIV positivity) or Hepatitis C (screening not required if no clinical suspicion)
* Evans Syndrome: positive direct Coombs with evidence of active hemolysis (elevated lactate dehydrogenase (LDH) or reticulocyte count not attributable to recent treatment or bleeding)
* Any Malignancy
* History of stem cell transplant or solid organ transplant
* aspartate aminotransferase (AST) or ALT >2 x upper limit of normal (ULN)
* Total bilirubin >1.5 × ULN
* Subjects with liver cirrhosis (as determined by the investigator)
* Creatinine >2.5 × ULN
* Known active or uncontrolled infections not responding to appropriate therapy
* On anticoagulation or anti-platelet agents
* Known thrombophilic risk factors. Exception: Subjects for whom the potential benefits of participating in the study outweigh the potential risks of thromboembolic events, as determined by the investigator.
* Baseline ophthalmic problems that may potentiate cataract development
* Impaired cardiac function, such as:

  * Known prolonged QTc, with corrected QTc >450 msec
  * Other clinically significant cardio-vascular disease (e.g., uncontrolled hypertension, history of labile hypertension),
  * History of known structural abnormalities (e.g. cardiomyopathy).
* History or current diagnosis of cardiac disease indicating significant risk of safety for patients participating in the study such as uncontrolled or significant cardiac disease, including any of the following:

  * Recent myocardial infarction (within last 6 months),
  * Uncontrolled congestive heart failure,
  * Unstable angina (within last 6 months),
  * Clinically significant (symptomatic) cardiac arrhythmias (e.g., sustained ventricular tachycardia, and clinically significant second or third degree AV block without a pacemaker.)
  * Long QT syndrome, family history of idiopathic sudden death, congenital long QT syndrome or additional risk factors for cardiac repolarization abnormality, as determined by the investigator.
* Known immediate or delayed hypersensitivity reaction to eltrombopag or its excipient.
* Pregnant, breastfeeding, or unwilling to practice birth control during participation in the study. Women of childbearing potential (have achieved menarche) must have a negative serum or urine pregnancy test and agree to use basic methods of contraception (if sexually active) or maintain abstinence for the duration of the study. Basic contraception methods include:

  * Total abstinence (when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception
  * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy), total hysterectomy, or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment
  * Male sterilization (at least 6 months prior to screening). The vasectomized male partner should be the sole partner for that subject
  * Barrier methods of contraception: Condom or Occlusive cap. For the UK: with spermicidal foam/gel/film/cream/ vaginal suppository
  * Use of oral, injected or implanted hormonal methods of contraception or placement of an intrauterine device (IUD) or intrauterine system (IUS), or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception. In case of use of oral contraception women should have been stable on the same pill for a minimum of 3 months before taking study treatment.
* Male patients who are sexually active and do not agree to abstinence or to use a condom during intercourse while taking eltrombopag, and for 7 days after stopping treatment.
* History of alcohol/drug abuse
* Presence of a medical condition that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data.
* Concurrent participation in an investigational study within 30 days prior to enrollment or within 5-half-lives of the investigational product, whichever is longer. Note: parallel enrollment in a non-therapeutic trial such as disease registry or biology study is permitted.

Other Eligibility Criteria Considerations All patients and/or their parents or legal guardians must sign a written informed consent (and assent when applicable)

* Patients and/or parents who are unable to read at a grade 2 level will be excluded from the patient-reported outcome component of the study, as will non-English speaking patients and/or parents when there is no availability of translated versions in their spoken language . They will not be excluded from all other aspects of the study

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 122 (Actual)
Dates: Start 2019-05-02 (Actual); Primary Completion 2024-04-17 (Actual); Study Completion 2025-02-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Grimes, MD, Principal Investigator — Baylor College of Medicine - Texas Children's Hospital
Locations (27):
- United States (27):
  - Children's of Alabama, Birmingham, Alabama
  - Phoenix CHildren's Hospital, Phoenix, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Children's Hospital of Orange County, Orange, California
  - UCSF Benioff Children's Hospital, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Florida College of Medicine, Gainesville, Florida
  - Alfac Cancer and Blood Disorder Center: Scottish Rite, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Riley Hospital for Children-Indiana University, Indianapolis, Indiana
  - Boston Children's Hospital, Boston, Massachusetts
  - Children's Hospital and Clinics of Minnesota, Minneapolis, Minnesota
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Columbia University Irving Medical Center, New York, New York
  - Weill Cornell Medical College, New York, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Nationwide Children's Hospital, Columbus, Ohio
  - Randall Children's Hospital, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Hasbro Children's Hospital, Providence, Rhode Island
  - St. Jude Children's Hospital, Memphis, Tennessee
  - Texas Children's Hospital, Houston, Texas
  - University of Wisconsin, Madison, Wisconsin

REFERENCES:
- [Derived] Shimano KA, Grimes AB, Kaicker S, Shah SJ, Gunn E, Bhat RV, Kochhar M, Rothman JA, Rose MJ, Briones M, Nakano TA, Lebensburger JD, Lambert MP, Fritch Lilla SA, Jesudas R, Lee-Miller CA, Thompson AA, Rifkin-Zenenberg S, Majumdar S, Crary SE, Hege K, Ford JB, Bies JJ, Fort J, Wynn TT, Hsieh L, Ruiz ME, Dinu B, Wong JMW, Kao PC, Kim TO, Arnold SD, Bennett CM, Despotovic JM, Klaassen RJ, Neufeld EJ, Neunert CE, London WB, Grace RF. Eltrombopag for Newly Diagnosed Pediatric Immune Thrombocytopenia Requiring Treatment: The PINES Randomized Clinical Trial. JAMA. 2025 Nov 25;334(20):1816-1826. doi: 10.1001/jama.2025.18168. PMID 41123939
- [Derived] Shimano KA, Grace RF, Despotovic JM, Neufeld EJ, Klaassen RJ, Bennett CM, Ma C, London WB, Neunert C. Phase 3 randomised trial of eltrombopag versus standard first-line pharmacological management for newly diagnosed immune thrombocytopaenia (ITP) in children: study protocol. BMJ Open. 2021 Aug 27;11(8):e044885. doi: 10.1136/bmjopen-2020-044885. PMID 34452956

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental: Eltrombopag: Patients ages 1 to <18 years with newly diagnosed primary ITP, platelets <30 x 10^9/L, requiring pharmacological treatment, but without severe bleeding or need for rapid rise in counts, randomized to receive the experimental therapy (eltrombopag).
- Comparator: Standard Therapy: Patients ages 1 to <18 years with newly diagnosed primary ITP, platelets <30 x 10^9/L, requiring pharmacological treatment, but without severe bleeding or need for rapid rise in counts, randomized to receive standard therapy (investigator choice of glucocorticoids, IVIg, anti-D immunoglobulin).
Period: Overall Study
Arm/Group | Experimental: Eltrombopag | Comparator: Standard Therapy
Started | 81 | 41
Completed | 78 | 40
Not Completed | 3 | 1
Not completed — patient retrospectively deemed ineligible (did not have primary ITP) | 2 | 0
Not completed — patient retrospectively deemed ineligible (Day 0 plt ct >30 x 10^9/L) | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental: Eltrombopag | Comparator: Standard Therapy | Total
Number analyzed (Participants) | 78 | 40 | 118
Age, Continuous [Median (Full Range); unit: years] | 7.9 [1.8 to 17.7] | 8.7 [1.1 to 17.2] | 8.2 [1.1 to 17.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 18 | 60
  Male | 36 | 22 | 58
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 11 | 26
  Not Hispanic or Latino | 56 | 27 | 83
  Unknown or Not Reported | 7 | 2 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 3 | 7
  White | 59 | 26 | 85
  More than one race | 3 | 1 | 4
  Unknown or Not Reported | 9 | 7 | 16

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With a Platelet Response
Description: To determine if the percentage of patients with a platelet response is significantly greater in patients with newly diagnosed ITP treated with eltrombopag than those treated with standard first-line treatments
Time Frame: 12 weeks
Population: This study included 118 pediatric patients (median age 8y, 49% male), 78 randomized to eltrombopag and 40 to standard therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: Eltrombopag | Comparator: Standard Therapy
Number analyzed (Participants) | 78 | 40
Participants | 52 | 14

2. Secondary Outcome: Bleeding Score
Description: Poor bleeding score (binary) at 1, 2, 3, 4 weeks, 12 weeks, and 1 year after study enrollment defined as World Health Organization (WHO) Bleeding Scale ≥ 2 or Modified Buchanan Scale ≥ 3
Time Frame: 1 year
Reporting Status: Not Posted

3. Secondary Outcome: Cumulative Number of Rescue Therapies Required
Description: The percentage of patients who received rescue therapy in the experimental (eltrombopag) arm vs the comparator (standard therapy) arm during the first 12 weeks of treatment
Time Frame: 12 weeks
Population: Patients who received >/= 1 dose of protocol-directed therapy were evaluable for secondary objectives.
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: Eltrombopag | Comparator: Standard Therapy
Number analyzed (Participants) | 78 | 39
Participants | 13 | 15

4. Secondary Outcome: Platelet Response Among Patients Requiring Rescue Therapy During Weeks 1-2 of Study
Description: Platelet response (binary), defined as ≥ 3 of 4 weeks with platelets >50 x109/L during weeks 6-12 of therapy, but patient required a rescue treatment during weeks 1-2 of study.
Time Frame: 12 weeks
Population: patient required a rescue treatment during weeks 1-2 of study.
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: Eltrombopag | Comparator: Standard Therapy
Number analyzed (Participants) | 6 | 2
Participants | 4 | 0

5. Secondary Outcome: Need for Treatment
Description: No further need for treatment (binary) after 12 weeks or 6 months of study
Time Frame: 6 months
Reporting Status: Not Posted

6. Secondary Outcome: Treatment Response
Description: Treatment response (binary endpoints) at 1 year defined as:
  * CR is defined as platelet count >/= 150 x 10^9/L
  * Primary Remission at 1 year is defined as CR at 1 year with no second-line agents required and >/= 3 months after discontinuing most recent platelet active medication
  * Disease resolution at 1 year is defined as complete response (CR) at 1 year >/= 3 months after discontinuing most recent platelet active medication. May have received a second-line therapy, excluding rituximab or splenectomy.
  * Disease stability at 1 year is defined as platelets >/= 50 x 10^9/L but <150 x 10^9/L >/= 3 months after discontinuing most recent platelet active medication.
Time Frame: 1 year
Reporting Status: Not Posted

7. Secondary Outcome: Number of 2nd Line Therapies
Description: Number of 2nd-line therapies in weeks 13-52
Time Frame: 52 weeks
Reporting Status: Not Posted

8. Secondary Outcome: Regulatory T-Cells
Description: Absolute change in percentage of CD4+25+Foxp3+ regulatory T cells from baseline at 12 weeks and 1 year
Time Frame: 1 year
Reporting Status: Not Posted

9. Secondary Outcome: KIT Scores
Description: Change in parent proxy-reported Kids ITP tool (KIT) overall scores from baseline at 1 week, 4 weeks, 12 weeks, and 1 year after study enrollment
Time Frame: 1 year
Reporting Status: Not Posted

10. Secondary Outcome: Hockenberry Fatigue Scale-Parent
Description: Total scale intensity ratings (continuous) from the Hockenberry Fatigue Scale-Parent (FS-P) at 1 week, 4 weeks, 12 weeks, and 1 year
Time Frame: 1 year
Reporting Status: Not Posted

11. Secondary Outcome: Blood Iron Values
Description: Serum iron, total iron binding capacity (TIBC), transferrin saturation, ferritin, mean corpuscular volume (MCV), and hemoglobin at 12 weeks, 6 months, and 1 year after study enrollment
Time Frame: 1 year
Reporting Status: Not Posted

12. Secondary Outcome: Safety Evaluations
Description: Safety evaluations as defined by:
  * Abnormal liver function tests (LFTs):
  ALT ≥ 3 x upper limit of normal (ULN) in patients with normal baseline ALT ≥ 3 x baseline or ≥ 5 x ULN (whichever is lower) in patients with abnormal baseline ALT ≥ 3 x ULN AND bilirubin ≥ 1.5 x ULN (>35% direct)
  * Incidence of adverse events
  * Incidence of serious adverse events
Time Frame: 1 year
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Time to Response
Description: Time to response (platelets >30x10^9/L, and at least 2-fold increase in the baseline count and absence of bleeding) (IWG definition)
Time Frame: 1 year
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Platelet-specific Endpoints
Description: Treatment response (platelets >30x10^9/L, and at least 2-fold increase in the baseline count and absence of bleeding) (IWG definition) at 12 weeks
Time Frame: 1 year
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Time to Platelet Count
Description: Time to platelet count >100x10^9/L and absence of bleeding (IWG definition)
Time Frame: 1 year
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Treatment Response
Description: Treatment response (platelet count >100x10^9/L and absence of bleeding) (IWG definition) at 12 weeks
Time Frame: 1 year
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Loss of Treatment Response
Description: Loss of treatment response (platelet count below 30x10^9/L, or less than 2-fold increase in the baseline count or bleeding) (IWG definition) at any time during the study period after achieving response during the first 12 weeks
Time Frame: 1 year
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Extreme Thrombocytosis
Description: Extreme thrombocytosis (platelets >1 x10^12/L)
Time Frame: 1 year
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Patient-reported Outcomes Endpoints
Description: Change in child self-reported and parent impact KIT scores from baseline at 1 week, 4 weeks, 12 weeks, and 1 year after study enrollment
Time Frame: 1 year
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Change in Hockenberry Fatigue
Description: Change in Hockenberry fatigue (FS-C, FS-A, FS-P) scores from baseline at 1 week, 4 weeks, 12 weeks, and 1 year after study enrollment
Time Frame: 1 year
Reporting Status: Not Posted

21. Other Pre Specified Outcome: Global Change Scale Scores
Description: Global Change Scale scores at 1 week, 4 weeks, 12 weeks, and 1 year after study enrollment
Time Frame: 1 year
Reporting Status: Not Posted

22. Other Pre Specified Outcome: Number of Hospitalizations
Description: Number of hospitalizations
Time Frame: 1 year
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 12 weeks (during which data was collected, and is now reported, in reference to the primary endpoint and/or primary outcome of the study -- proportion of patients achieving a durable platelet response of at least 3 of 4 platelet counts over 50 x10^9/L without rescue therapy during weeks 6-12 of study)
Description: Adverse Events of Grade 3 or higher during the first 12 weeks on study (as defined by the CTCAE v5.0) are reported for all patients who received at least one dose of treatment (n=117)
Arm/Group | Experimental: Eltrombopag | Comparator: Standard Therapy
All-Cause Mortality (participants affected / at risk) | 0/78 | 0/39
Serious Adverse Events (participants affected / at risk) | 6/78 | 3/39
Other Adverse Events (participants affected / at risk) | 8/78 | 3/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: Eltrombopag (N=78) | Comparator: Standard Therapy (N=39)
Hemotympanum (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hematoma (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Urinary Tract Infection (Renal and urinary disorders) | 1 (1) | 0 (0)
Allergic Reaction (Immune system disorders) | 0 (0) | 1 (1)
Epistaxis (Ear and labyrinth disorders) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: Eltrombopag (N=78) | Comparator: Standard Therapy (N=39)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Epistaxis (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 3 (3)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-06-26): https://cdn.clinicaltrials.gov/large-docs/37/NCT03939637/Prot_SAP_000.pdf